CLINICAL TRIAL: NCT07256600
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Bioequivalence After Administration of "DWJ1445" and "DWC202506" in Healthy Adults
Brief Title: PK and Safety Comparison of DWJ445 and DWC202506 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1445102
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(RT) (Experimental): 35 subjects, Cross-over, Single dose DWC202506 on period 1, Single dose of DWJ1445 on period 2
  Interventions: Drug: DWJ1445; Drug: DWC202506
- B(TR) (Experimental): 35 subjects, Cross-over, Single dose DWJ1445 on period 1, Single dose of DWC202506 on period 2
  Interventions: Drug: DWJ1445; Drug: DWC202506

INTERVENTIONS:
Drug: DWJ1445 — 1 tablet, Orally
Drug: DWC202506 — 1 tablet, Orally

SUMMARY:
A bioequivalence study comparing DWJ1445 and DWC202506 in healthy adults

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, 2-treatment, 2-period, crossover, bioequivalence study conducted under fasting conditions to compare and evaluate the pharmacokinetics and safety of DWJ1445 and DWC202506 in healthy adult volunteers. Participants will receive both study drugs in separate periods, with a washout interval between administrations. The study aims to assess PK parameters and monitor safety through clinical evaluations and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a body mass index (BMI) between 18 and 30 kg/m²
* Subjects without any clinically significant congenital or chronic disease, and with no pathological findings based on medical examination
* Subjects who agree to use a medically acceptable method of contraception

Exclusion Criteria:

* Subjects who have participated in a bioequivalence or other clinical trial and received an investigational product within 6 months prior to the first dose
* Subjects with a history of gastrointestinal surgery that may affect drug absorption
* Subjects with a clinically significant history of psychiatric illness Female subjects who are pregnant, suspected of being pregnant, or currently breastfeeding

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-11-14 (Actual); Primary Completion 2025-11-23 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-24 hours
  Area under the plasma drug concentration-time curve [AUCt] of DWJ1445 and DWC202506
Maximum plasma concentration [Cmax] | 0-24 hours
  Maximum plasma concentration [Cmax] of DWJ1445 and DWC202506

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity | 0-24 hours
  Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] of DWJ1445 and DWC202506
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-24 hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] of DWJ1445 and DWC202506
Time of peak concentration [Tmax] | 0-24 hours
  Time of peak concentration [Tmax] of Amoxicillin & Clavulanic acid of DWJ1445 and DWC202506
Terminal phase of half-life [t1/2] | 0-24 hours
  Terminal phase of half-life of DWJ1445 and DWC202506

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No